CLINICAL TRIAL: NCT07372326
Title: A Study on the Effect of Electronic Moxibustion Based on Ziwu Liuzhu in Treating Constipation in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-2025-055
Record Dates: First submitted 2025-12-11; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Stroke Patients With Constipation
Keywords: cerebral hemorrhage; constipation; midnight-midday ebb flow; electronic moxibustion
MeSH Terms: conditions — Cerebral Hemorrhage; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional nursing methods for treating constipation after stroke (No Intervention): (1) Basic treatment includes drug therapy: oral and intravenous medications are administered based on the principles of "controlling blood pressure, blood sugar, and anti-platelet aggregation". (2) Psychological care. Provide psychological and comfort care for the patients to enable them to receive treatment in a comfortable and hospitable environment. (3) Dietary care. Adopt a light diet and increase intake of low-fat, high-fiber, high-vitamin, and high-protein foods. (4) Rehabilitation exercises: bedpan training, abdominal massage, etc.
- Electro-acupuncture therapy under the guidance of the theory of meridian flow (Experimental): The intervention group C patients were given electronic moxibustion therapy based on the theory of Ziwen Liuzhun (midnight to dawn) under the premise of the control group B. According to the theory of Ziwen Liuzhun, the hour of Ba (05:00 - 07:00) is the time when the large intestine meridian is in charge, and at this time, the blood and qi of the large intestine are abundant, which is most conducive to excretion. The hour of Chen (07:00 - 09:00) is the time when the stomach meridian is in charge, and at this time, the qi of the stomach meridian is vigorous, which is most conducive to regulating the connection between the stomach and the spleen. Based on the specific conditions of each patient, moxibustion treatment was given at the corresponding hour. The specific moxibustion therapy was the same as that of the control group. The intervention lasted for 2 weeks.
  Interventions: Device: An electronic moxibustion device under the guidance of the Yuziuyouluo theory
- electronic moxibustion (Experimental): The intervention group B added electronic moxibustion to the treatment of group A: Assist the patient to assume the supine position, aim at the moxibustion areas around the navel (Shenque, Guanyuan, Qihai, Xiaquan, Tianqiu), and use electronic moxibustion therapy (Production License No. 20180137 of Su Food and Drug Administration). The distance from the skin was 5 to 10 cm, and each area was moxibustion for 30 minutes. During the moxibustion process, ask the patient if there is any discomfort, observe the patient's skin condition, and assist the patient to put on clothes and take a comfortable lying position after the treatment.
  Interventions: Device: Electronic moxibustion instrument

INTERVENTIONS:
Device: Electronic moxibustion instrument — The intervention group B added electronic moxibustion to the treatment of group A: Assist the patient to assume the supine position, aim at the moxibustion areas around the navel (Shenque, Guanyuan, Qihai, Xiaowan, Tianqiu), and use electronic moxibustion therapy (Production License No. 20180137 of Su Food and Drug Administration). The distance from the skin is 5 to 10 cm, and each area is moxibustion for 30 minutes. During the moxibustion process, ask the patient if there is any discomfort, observe the patient's skin condition, and assist the patient to put on clothes and take a comfortable lying position after the treatment.
  Arms: electronic moxibustion
Device: An electronic moxibustion device under the guidance of the Yuziuyouluo theory — The intervention group C patients were given electronic moxibustion therapy based on the theory of Ziwen Liuzhun (midnight to dawn) under the premise of the control group B. According to the theory of Ziwen Liuzhun, the hour of Ba (05:00 - 07:00) is the time when the large intestine meridian is in charge, and at this time, the blood and qi of the large intestine are abundant, which is most conducive to excretion. The hour of Chen (07:00 - 09:00) is the time when the stomach meridian is in charge, and at this time, the qi of the stomach meridian is vigorous, which is most conducive to regulating the connection between the stomach and the spleen. Based on the specific conditions of each patient, moxibustion treatment was given at the corresponding hour. The specific moxibustion therapy was the same as that of the control group. The intervention lasted for 2 weeks.
  Arms: Electro-acupuncture therapy under the guidance of the theory of meridian flow

SUMMARY:
This study aims to explore the application effect of Ziwu Liuzhu electronic moxibustion combined with auricular points on constipation in stroke patients through clinical controlled trials, as well as the advantages over using electronic moxibustion alone.

DETAILED DESCRIPTION:
This study aims to explore the application effect of Ziwu Liuzhu electronic moxibustion combined with auricular points on constipation in stroke patients through clinical controlled trials, as well as the advantages over using electronic moxibustion alone. It provides new explorations, new ideas and new methods for the effective clinical care of constipation in stroke patients, and offers theoretical and guiding basis for the application and promotion of electronic moxibustion.

ELIGIBILITY:
Inclusion criteria:

1. Meets the diagnostic criteria of both Western medicine and traditional Chinese medicine, and has not undergone surgery or other internal medical treatments, with the occurrence of constipation;
2. The condition is stable, without severe clinical complications;
3. Can accept moxibustion treatment, and the local skin is undamaged;
4. Those who agree to participate in this study and sign the informed consent form.

Exclusion criteria:

1. Digestive tract disorders, such as intestinal polyps, tuberculosis, and tumors. Irritable bowel syndrome or constipation secondary to organic diseases (such as endocrine, metabolic or post-operative diseases); abdominal aneurysm, hepatosplenomegaly, or severe cardiovascular, liver, kidney or mental disorders and coagulation disorders.
2. The patient had constipation before the stroke.
3. The patient withdrew from the study due to other reasons during the course of the study.

Dropout criteria and termination criteria:

1. Patients who have not received the prescribed treatment and whose therapeutic effect cannot be determined;
2. Patients who experience serious adverse events or complications and are not suitable to continue the treatment and thus the trial is terminated;
3. Patients with poor compliance, who withdraw from the treatment during the course of the trial, or who use treatment methods prohibited by this protocol concurrently, or who change the treatment method halfway on their own.

Note: For any patient meeting any of the above criteria 1, they will be handled as a dropout case.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The first time of defecation | The timing of the intervention starts from the moment it begins until the first successful defecation occurs, and is recorded in hours (h).

SECONDARY OUTCOMES:
Clinical Symptom Score Scale (CCS) | An assessment was conducted before the experimental intervention, on the 7th day of the intervention, and after the completion of the intervention.
  CCSis mainly used to assess the severity of constipation and has good reliability and validity. It is widely used in clinical trial evaluations. The items involved all match the items of the Rome IV standard. Except for one item with a score range of 0-7, the score range of all other items is 0-4. The higher the total score, the more severe the constipation.

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Zhejiang University, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No